CLINICAL TRIAL: NCT04328467
Title: Pre-exposure Prophylaxis for SARS-Coronavirus-2: A Pragmatic Randomized Clinical Trial
Brief Title: Pre-exposure Prophylaxis for SARS-Coronavirus-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED-2020-28720
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: COVID-19; Corona Virus Infection; ARDS; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Distress Syndrome | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intervention Once Weekly (Experimental): 400 mg orally once, followed by 400mg 6 to 8 hours later, thereafter 400mg weekly for the duration of follow up, up to 12 weeks
  Interventions: Drug: Hydroxychloroquine
- Intervention Twice Weekly (Experimental): 400mg orally once, followed by 400mg 6 to 8 hours later, thereafter 400mg twice weekly for the duration of follow up, up to 12 weeks
  Interventions: Drug: Hydroxychloroquine
- Control Group (Placebo Comparator): Placebo 2 tabs once, followed by 2 tabs 6 to 8 hours later, thereafter two tabs weekly or twice weekly for the duration of follow up, up to 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine; 200mg tablet; oral
  Other Names: Plaquenil
  Arms: Intervention Once Weekly; Intervention Twice Weekly
Other: Placebo — Placebo; tablet; oral
  Arms: Control Group

SUMMARY:
Objective: To determine if pre-exposure prophylaxis with hydroxychloroquine is effective for the prevention of COVID-19 disease.

DETAILED DESCRIPTION:
The current standard of care is observation and quarantine after exposure to COVID-19. There is no approved treatment or prophylaxis for COVID-19.

As of March 6, 2020, the CDC estimates that the transmission of SARS-CoV2 after a U.S. household close contract is 10.5% (95%CI, 2.9 to 31.4%). Among all close contacts, the SARS-CoV2 transmission rate is estimated at 0.45% (95%CI, 0.12 to 1.6%) by the CDC. These estimates are based on monitoring of travel-associated COVID19 cases. Conversely, in a setting with community transmission, the secondary attack rate in China was 35% (95%CI, 27-44%) based on 48 transmissions among 137 persons in 9 index patients.

Chloroquine or Hydroxychloroquine may have antiviral effects against SARS-COV2 which may prevent COVID-19 disease or reduce disease severity. It is not known at what dosing hydroxychloroquine may be effective for pre-exposure prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

- A healthcare worker at high risk for COVID-19 exposure (defined below):

* Persons primarily working in emergency departments (physicians, nurses, ancillary staff, triage personnel)
* Persons primarily working in intensive care units (physicians, nurses, ancillary staff, respiratory therapists)
* Persons performing aerosol generating procedures (i.e. anesthesiologists, nurse anesthetists (CRNAs)
* First responders (i.e. EMTs, paramedics)

Exclusion Criteria:

* Active COVID-19 disease
* Prior COVID-19 disease
* Current fever, cough, shortness of breath
* Allergy to chloroquine or hydroxychloroquine
* Prior retinal eye disease
* Known Chronic Kidney disease, Stage 4 or 5 or dialysis
* Known glucose-6 phosphate dehydrogenase (G-6-PD) deficiency
* Weight <40 kg
* Prolonged QT syndrome
* Current use of hydroxychloroquine, chloroquine, or cardiac medicines of flecainide, amiodarone, digoxin, procainamide, or propafenone
* Current use of medications with known significant drug-drug interactions: artemether, lumefantrine, mefloquine, tamoxifen, or methotrexate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1483 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radha Rajasingham, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Nationwide Enrollment via Internet, please email: covid19@umn.edu, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rajasingham R, Bangdiwala AS, Nicol MR, Skipper CP, Pastick KA, Axelrod ML, Pullen MF, Nascene AA, Williams DA, Engen NW, Okafor EC, Rini BI, Mayer IA, McDonald EG, Lee TC, Li P, MacKenzie LJ, Balko JM, Dunlop SJ, Hullsiek KH, Boulware DR, Lofgren SM; COVID PREP team. Hydroxychloroquine as Pre-exposure Prophylaxis for Coronavirus Disease 2019 (COVID-19) in Healthcare Workers: A Randomized Trial. Clin Infect Dis. 2021 Jun 1;72(11):e835-e843. doi: 10.1093/cid/ciaa1571. PMID 33068425
- [Derived] Lofgren SM, Nicol MR, Bangdiwala AS, Pastick KA, Okafor EC, Skipper CP, Pullen MF, Engen NW, Abassi M, Williams DA, Nascene AA, Axelrod ML, Lother SA, MacKenzie LJ, Drobot G, Marten N, Cheng MP, Zarychanski R, Schwartz IS, Silverman M, Chagla Z, Kelly LE, McDonald EG, Lee TC, Hullsiek KH, Boulware DR, Rajasingham R. Safety of Hydroxychloroquine Among Outpatient Clinical Trial Participants for COVID-19. Open Forum Infect Dis. 2020 Oct 19;7(11):ofaa500. doi: 10.1093/ofid/ofaa500. eCollection 2020 Nov. PMID 33204764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Started | 494 | 495 | 494
Completed | 490 | 493 | 493
Not Completed | 4 | 2 | 1
Not completed — Did not meet inclusion criteria after randomization | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group | Total
Number analyzed (Participants) | 494 | 495 | 494 | 1483
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 42 [35 to 49] | 41 [35 to 49] | 40 [34 to 48] | 41 [35 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 261 | 258 | 241 | 760
  Male | 233 | 237 | 253 | 723
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 431 | 421 | 419 | 1271
  Black of African | 5 | 5 | 10 | 20
  Asian | 23 | 23 | 29 | 75
  Native Hawaiian or Pacific Islander | 0 | 1 | 1 | 2
  Hispanic or Latino | 18 | 22 | 18 | 58
  Native American or Alaska Native | 4 | 7 | 8 | 19
  Middle Eastern | 6 | 5 | 4 | 15
  South Asian | 17 | 18 | 12 | 47
  Other | 3 | 1 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 493 | 494 | 493 | 1480
  Canada | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: COVID-19-free Survival
Description: Outcome reported as the number of participants in each arm who are COVID-19-free at the end of study treatment.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Number analyzed (Participants) | 494 | 495 | 494
Participants | 464 | 468 | 454

2. Secondary Outcome: Number of Confirmed SARS-CoV-2 Detection
Description: Outcome reported as the number of participants in each arm who have a confirmed SARS-CoV-2 infection during study treatment.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Number analyzed (Participants) | 494 | 495 | 494
Participants | 29 | 29 | 39

3. Secondary Outcome: Incidence of Possible COVID-19 Symptoms
Description: Outcome reported as the count of participants in each arm who report COVID-19-related symptoms during study treatment.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Number analyzed (Participants) | 494 | 495 | 494
Participants | 29 | 28 | 38

4. Secondary Outcome: Incidence of All-cause Study Medicine Discontinuation
Description: Outcome reported as the count of participants in each arm who discontinue study medication use for any reason during treatment.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Number analyzed (Participants) | 494 | 495 | 494
Participants | 119 | 158 | 133

5. Secondary Outcome: Ordinal Scale of COVID-19 Disease Maximum Severity if COVID-19 Diagnosed at Study End
Description: Participants will self-report COVID-19 status on an ordinal scale as follows: No illness (score=1), Illness with outpatient observation (score=2), Hospitalization (or post-hospital discharge) (score=3), or Hospitalization with ICU stay or death (score=4). Possible scores range from 1-4 with higher scores indicating greater disease severity.
Time Frame: up to 12 weeks
Population: Measure was only collected for one participant in the twice-weekly intervention group and one participant in the control group. No participants in the once-weekly intervention group were sampled for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Number analyzed (Participants) | 0 | 1 | 1
score on a scale |  | 1 (NA) — Only one data point was collected, therefore a measure of dispersion could not be calculated. | 1 (NA) — Only one data point was collected, therefore a measure of dispersion could not be calculated.

6. Secondary Outcome: Incidence of Hospitalization for COVID-19 or Death
Description: Outcome reported as the number of participants in each arm who are hospitalized or expire due to COVID-19 during study treatment.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Number analyzed (Participants) | 494 | 495 | 494
Participants | 3 | 8 | 9

7. Secondary Outcome: Incidence of Possible Study Medication-related Side Effects
Description: Outcome reported as the number of participants in each arm who experience possible medication-related side effects during study treatment.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
Number analyzed (Participants) | 494 | 495 | 494
Participants | 148 | 168 | 100

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Arm/Group | Intervention Once Weekly | Intervention Twice Weekly | Control Group
All-Cause Mortality (participants affected / at risk) | 0/494 | 0/495 | 0/494
Serious Adverse Events (participants affected / at risk) | 3/494 | 6/495 | 8/494
Other Adverse Events (participants affected / at risk) | 0/494 | 0/495 | 0/494
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Once Weekly (N=494) | Intervention Twice Weekly (N=495) | Control Group (N=494)
Hysteroscopy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Elective Coronary Angiogram (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Gall Bladder Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Heart Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sarcoidosis Biopsy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Other Not Specified (General disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT04328467/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04328467/ICF_001.pdf